## **Study Title**

Effect of Patient Information Leaflet on working pattern and patient satisfaction level in a busy Indian day care operative theatre complex

## **Investigators**

## Dr. Sumitra Bakshi

MD, DNB (Anaesthesiology)

Professor

Department of Anaesthesia, Critical Care and Pain

# Dr. Amit Raja Panigrahi

Post-graduate Student,
Department of Anaesthesia, Critical Care and Pain

### Dr. Akash Tambule

Post-graduate Student,
Department of Anaesthesia, Critical Care and Pain

#### Dr. Prathamesh Pai

M.S.

Professor

Department of Surgical Oncology

# **Institution**

Tata Memorial Hospital, Mumbai-400 012

# **Table of Contents**

- 1. Study summary
- 2. Introduction
- 3. Aims and objectives
- 4. Inclusion and exclusion criteria
- 5. Material and methods
- 6. Measurements
- 7. Statistical analysis
- 8. References

**Annexure form 2.1** 

Annexure form 2.2

Study title: Effect of Patient Information Leaflet on working pattern and patient

satisfaction level in a busy Indian day care operative theatre complex

Investigator: Dr Sumitra Bakshi, Dr Amit Raja Panigrahi, Dr Akash Tambule,

Dr Prathamesh Pai

Study Site: Department of Anaesthesia, Critical Care and Pain, Tata Memorial Hospital,

Parel, Mumbai 400 012.

**INTRODUCTION:** 

Patient Information is one of the key determinants of patient satisfaction. Adequate

information about the disease condition, treatment plan, waiting times and 'what to do next'

affects patients' overall satisfaction level. Good quality information not only reduces patient

anxiety and stress but also reduces unreasonable expectations and misperceptions. Patient

satisfaction has always remained an important and commonly used indicator for measuring

the quality in health care.

In the recent years there is a gradual upward trend in day care surgeries all across the

globe; an estimated 83% of the surgeries in the United States being performed on an

ambulatory basis<sup>1</sup>. In India, about 20 percent of all surgical procedures are performed on

outpatients. It is estimated that by 2020, 75 percent of all surgical operations in India will be

carried out in ambulatory surgery centers <sup>2</sup>. The increasing trend of ambulatory surgeries has

emerged from advances in anesthesia and surgical techniques. Patient information and

effective communication is critical in these surgeries especially the ones that need General

Anesthesia. Provision of information is one of the mainstays of effective day surgery

management. This needs to cover not only what to do preoperatively and postoperatively, but

also what will happen on the day of surgery. There are several ways of providing information

like written information, using a video, over telephone or by patient interviews before and

Version1

after surgery. Verbal information alone is inadequate and must be reinforced with well-

presented printed material<sup>3</sup>.

Tata Memorial hospital is a premier tertiary level cancer hospital in India. Around 140-

150 patients undergo minor surgical procedures (diagnostic and therapeutic) in our hospital's

Minor OT complex every day. About 30-40% of surgeries belong to the Head & Neck region

alone. About 40-50% of these surgeries are done under General Anaesthesia. At present the

communication with patients in the busy outpatient department is mainly verbal. Due to time

constrains, lack of a responsible attendant with the patient, important information with respect

to the day care procedure is often not effectively delivered. This leads to patients not following

instruction adequately with respect to starvation, medications to be taken on the day of the

procedure and also not carrying all essential documents. This leads to delays, rescheduling of

cases and rarely postponement of procedures.

Does an information leaflet provide an effective way of communication in the peri-

procedure period? Will it help in better information delivery and hence reduce the number of

avoidable postponements and delay. And does this translate to better patient satisfaction is want

this study aims to see. The study is restricted to patients undergoing Head & Neck procedures

under General Anaesthesia, as they form the major bulk of patients in our minor OT complex

and for logistic reasons to start with a defined group of patients.

**AIMS AND OBJECTIVES:** 

1. To reduce postponement of cases due to lack of information to patients in the pre-

operative period

2. To compare satisfaction levels between patients, pre and post introduction of

information leaflet

Version1

**Primary end point:** 

To reduce postponement of cases due to lack of information to patients in the pre-operative

period

Co Primary end point:

To compare satisfaction levels between patients, pre and post introduction of information

leaflet.

**Design of the study:** Pre and post interventional model

**INCLUSION CRITERIA:** 

All adult patients (> 18yrs), ASA I-III, undergoing elective therapeutic/diagnostic Head &

Neck surgeries under General Anaesthesia in the Minor OT complex and discharged on the

same day will be included. The surgeries will include Head & Neck surgeries like DL

scopies, laser surgeries, EUA, excision biopsies etc.

**EXCLUSION CRITERIA:** 

1. Patients refusing to take part in study

2. Patients undergoing emergency surgeries

3. ASA IV patients, or high risk patients planned for admission

4. Admitted patients for minor OT procedure

**5.** Patients not getting the Information leaflet due to any reason (in 2<sup>nd</sup> half of study)

**6.** Patient and his attendant, both illiterate

Version1

MATERIAL AND METHODS

After Institutional Review Board approval, all adult patients meeting inclusion criteria

and undergoing surgeries in the Minor OT complex during a 6 month period will be enrolled

in the study. The study will be done in two parts.

In the First half of study- planned over 2 months (Nov-Dec), feedback forms will be

collected from patients at the end of minor OT procedure (Annexure 2.1) All patients,

meeting inclusion criteria, at the end of the procedure prior to discharge from the minor OT

will be explained about the study and they shall be given a feedback form to be filled and

submitted. Also the number of postponement or rescheduling of cases will be noted.

Postponement or rescheduling of case is defined as an event when the patient who is

called for his turn in minor OT is deferred for any amount of time in account of starvation not

adequate, investigations not brought, medications not taken as prescribed. Any postponement

in view of awaiting opinion form senior consultant, special equipment or any investigations

called in view of patients clinical conditions which was not anticipated in the OPD by the

surgical colleague, or due to lack of OT time will not be included.

After the initial collection of feedback over 2 months, the patient information leaflet (PIL) will

be handed over to all patients planned for procedure in the minor OT complex (Second half of

study). This leaflet will be handed over by the attending doctor in the Head neck OPD. The

checklist pertaining to counselling at the Head neck OPD will be ticked after they are carried

out. The patient will be instructed to read leaflet carefully and carry the leaflet on the day of

Minor OT procedure. In the minor OT the discharge checklist in the PIL would be carried out

by all concerned including the surgical, anesthesia and nursing team. A period of 1 month (Jan)

will be allowed to streamline the use of patient information leaflet.

Version1

In the subsequent 2 months, Feb - Mar, the impact of use of PIL will be assessed. Firstly

by noting the number of postponement or rescheduling of cases. In addition all patients meeting

inclusion criteria will be given the feedback form (Annexure 2.2) at the end of their procedure

in minor OT.

For patients coming to minor OT without a patient information leaflet- one would ascertain if

the leaflet was handed in OPD and not brought to minor OT or if the leaflet was not handed at

all. The numbers of such misses will be recorded. Patients who did not get the leaflet in the

OPD will be excluded from study.

Sample size calculation:

For our preliminary review of postponement rate as defined in our study is around 20%. We

aim for a reduction of such postponement by 50%. Group sample sizes of 199 in group 1 and

199 in group 2 achieve 80.007% power to detect a difference between the group proportions

of -0.1000. The proportion in group 1 (the treatment group) is assumed to be 0.2000 under

the null hypothesis and 0.1000 under the alternative hypothesis. The proportion in group 2

(the control group) is 0.2000. The test statistic used is the two-sided Z-Test with pooled

variance. The significance level of the test is 0.0500. Considering a 20% loss to follow up

from OPD to minor OT, the sample size needed is 480 patients. On an average at least 250

patients of head neck patients undergo procedure under general anesthesia, per month (12-15

patients /day x 20 working days). With due consideration of our inclusion criteria, a two

month recruitment period pre and post intervention should be adequate.

**MEASUREMENTS** 

Version1

- No. of cases postponed pre and post introduction of the leaflet and reasons behind them
- Primary data collected will be patient satisfaction levels after the procedure (both pre and post PIL) on a 5 point Likert scale (Ranging from very poor = 0 to Excellent = 4)
- No of patients who did not receive the patient information leaflet in the OPD
- No of patients who received the PIL but did not get it along to the minor OT

#### STATISTICAL ANALYSIS

All Data will be analyzed using SPSS software. Likert scores will be treated as ordinal data. Proportions will be compared using chi square analysis. Additionally Multivariate logistic regression analysis will be used to assess the contribution of possible covariates, including age sex and patient knowledge on patient satisfaction. For all data P-value < 0.05 will be considered as statistical significant.

#### **REFERENCES:**

- 1. Beverly K. Philip MD, Day Care Surgery: The United States Model of Health Care IAAS Journal/17.4/PHILIP17.4.pdf
- 2. Emerging Trends in Healthcare A Journey from Bench to Bedside 17 February 2011;KPMG/ASSOCHAM
- 3. Jarrett, P. E. M, Day care surgery ;European Journal Of Anaesthesiology November 2001 Volume 18 Issue p 32–35
- 4. Shah U, Wong DT, Wong JPatient satisfaction and positive patient outcomes in ambulatory anesthesia 9 April 2015 Volume 2015:2 Pages 29—37 dovepress.com

# Annexure 2.1

Version1 Dtd. 12/08/2016 You are invited to take part in this study & help us improve the quality of services provided to you. Your participation is completely voluntary & it will not alter the treatment given to the patient in any way. Please base your answers on today's experience at this MINOR OT COMPLEX. Just mark the option which the patient thinks is correct.

| 1. Patients a | ige | Gender | | | |
|---|---|---|---|---|---|
| 2. Education | n: Illiterate/ | school/ graduate | / post gra | duate (please ti | ck patients highest qualification) |
| 3. Are you fi | lling this qu | uestionnaire for $\Box$ | self or 🗆 | on behalf of the | patient?, |
| If Yes (pleas | e tick your l | highest qualificati | on) Educa | ation Illiterate/s | school/ graduate/ post graduate |
| 4. Is this you | ır first visit | to this Minor OT o | complex? | Yes | No |
| If "No" when was the last time you came here? | | | | | |
| 5. Were you<br>eat/drink)? | adequately | y informed with re | egard to t | he fasting proce | edure, pre-surgery (What to |
| Yes | No | Not sure | | | |
| 6. Were you<br>the procedu | | about any tests (b | lood tests | s, ecg, scans,x-ra | ey etc.) that were necessary before |
| Yes | No | Not sure | | | |
| 7. If you tak<br>or to avoid | • | _ | oasis, wer | e you informed | about which medicines to continue |
| Yes | No | Not sure | | | |
| • | | - | | | action about your treatment reatment & follow up) |
| Yes | No | Not sure | | | |
| 9. How was surgery? | your overal | ll satisfaction with | respect t | to the informati | on you were provided <u>before</u> the |
| Excellent | Very goo | d Good | Poor | Very Poor | |
| 10. How wa surgery? | s your over | all satisfaction wit | th respect | to the informat | tion you were provided <u>after</u> the |
| Excellent | Very goo | d Good | Poor | Very Poor | |

# Annexure 2.2

You are invited to take part in this study & help us improve the quality of services provided to you. Your participation is completely voluntary & it will not alter the treatment given to the patient in any way. Please base your answers on today's experience at this MINOR OT COMPLEX. Just mark the option which the patient thinks is correct.

| 1. Patients a | ge | Gender | | | | |
|---|---|---|---|---|---|---|
| 2. Education Illiterate/ school/ graduate/ post graduate (please tick patient's highest qualification) | | | | | | |
| | _ | uestionnaire for<br>ducation Illiterate | | | - | olease tick your |
| • | | to this Minor OT ollow | • | | No | |
| 5. Were you<br>eat/drink)? | adequately | y informed with r | egard to tl | ne fasting proce | edure, pre-surge | ry (What to |
| Yes | No | Not sure | | | | |
| the procedu | | about any tests (b<br>Not sure | lood tests | , ecg, scans,x-ra | ay etc.) that were | e necessary before |
| . If you take any medicine on a regular basis, were you informed about which medicines to continue r to avoid on the day of surgery?<br>es No Not sure | | | | | | |
| | | igh information a<br>ct the result of to<br>Not sure | | | • | |
| 9. Have you<br>Yes | received ar<br>No | ny Information lea | aflet at the | e OPD? | | |
| lf "yes "have<br>Yes | you read t<br>No | the leaflet? | | | | |
| lf "yes "have<br>Yes | e you under<br>No | rstood the inform | ation prov | rided in the leaf | flet? | |
| | | n about the leafle<br>erage Bad Very B | | | | |
| • | | nend this leaflet to<br>will Recommen | | /recommend r | eluctantly/ not r | ecommend at all |
| | s your over | all satisfaction wi | th respect | to the informa | tion you were pr | ovided <u>before</u> the |
| surgery?<br>Excellent | Very goo | d Good | Poor | Very Poor | | |
| 13. How was | s your over | all satisfaction wi | th respect | to the informa | tion you were pr | ovided <u>after</u> the |
| Excellent | Very goo | d Good | Poor | Very Poor | | |
| Version1 | | | | | | |